CLINICAL TRIAL: NCT01693484
Title: Application of Indocyanine Green Angiography for Closed Operative Calcaneus Fractures Requiring Extensile Lateral Incision
Brief Title: Application of Indocyanine Green Angiography for Closed Operative Calcaneus Fractures
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Resource availability
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Todd Jaeblon, Associate Professor of Orthopaedic Surgery; Associate Director of Othopaedic Trauma, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICGVA-OS CALCIS 2012
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Fractures, Comminuted; Surgical Wound Dehiscence; Necrosis
Keywords: Calcaneus; Fracture; Indocyanine Green; Angiography; Open Reduction and Internal Fixation
MeSH Terms: conditions — Fractures, Comminuted; Surgical Wound Dehiscence; Necrosis; Fractures, Bone | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICG administered (Experimental): The ICG dose (10 mg/4cc per image capture) will be administered in its entirety via push injection through IV access established for standard surgical procedure, followed by 10 cc Normal Saline bolus. This ICG dose will be administered twice, 1X prior to anesthesia, and 1X after the tourniquet on operative extremity has been removed for at least 15 minutes.
  Interventions: Drug: ICG (Indocyanine Green)

INTERVENTIONS:
Drug: ICG (Indocyanine Green) — Diagnostic drug used for visualisation of blood perfusion in various tissues.Administered intravenously, 2X: 1X prior to anesthesia, and 1X after tourniquet on operative extremity has been released for at least 15 minutes. When excited by laser light source, it subsequently emits at a near infrared frequency.
  Other Names: NDC # 75874-0701-25

SUMMARY:
Researchers in the Orthopaedic surgery department at LSU Medical Center-Shreveport hope to learn if patterns of blood-flow around the incision site of patients undergoing surgery for heel-bone fractures can help predict whether complications will arise after a specific type of operation.The goals of this research study are to effectively answer as many of the following research questions as possible:

1. Can a drug normally used to evaluate adequate blood flow in plastic surgery and tissue transfer be used to identify altered patterns of blood flow at the operative site of Calcaneus fractures, when compared to the uninjured extremity?
2. Are changes in blood flow identifiable at the operative site post operatively?
3. Are there certain patterns of blood flow present preoperatively or postoperatively that can predict wound complication?
4. Can certain patterns of blood flow predict the location of slough or dehiscence after surgery?
5. Does the incision site and its proximity to specific patterns of blood flow possibly predict wound complication?

The hypothesis is that the study drug will show a correlation between certain patterns of blood flow and whatever post-operative complications may arise.

DETAILED DESCRIPTION:
Fractures of the calcaneus comprise 2% of all adult fractures. These fractures make up 60% of all tarsal injuries, the majority of which are closed, displaced intra-articular fractures. Despite the injury's prevalence, dispute over the appropriate method of treatment remains ongoing. Several studies have shown that an open, surgical approach is superior to either a non-surgical or percutaneous approach with regard to restoring proper alignment and structure of the hindfoot, depending on the severity of the displacement, and provided that certain patient conditions do not preclude surgery. Adequately restoring hindfoot structure is paramount to good clinical outcome; not only is proper alignment integral for fully recovering physiological functionality, but also in preventing further complications such as subtalar arthritis that present commonly in malunited calcaneal fractures.

Though literature may show that open reduction and internal fixation (ORIF) techniques provide a better long term outcome of severely displaced intra-articular fractures, proponents of both non surgical and percutaneous approaches argue that the superiority of the outcome may be mitigated by the fact that open surgical procedures are laden post operatively with numerous wound complications. These complications include, but are not limited to, both deep and superficial infections resulting in slough, dehiscence, necrosis, and erythema in and around the surgical site. Managing infections of the surrounding soft tissue and vasculature of the calcaneus following operative treatment indeed seems to present a great challenge to treating physicians, with wound healing complications present in 2-25% of cases.

A necessity for surgical wound repair is adequately vascularized tissue, which can be difficult to come by during closure of the wound due to the undermining and displacement of soft tissue during surgery. Sufficiently perfused soft tissue can also be difficult to differentiate from tissues that are inadequately vascular based on traditional clinical criteria such as color, warmth, and dermal bleeding. The degree of this avascularity can depend on many factors relating to the patient, necessitating studies be conducted identifying what factors place a prospective patient at a higher risk for developing wound healing problems post operatively. Studies of this nature thus far have noted that factors such as age, sex, height, weight, Bohler's angle, tobacco usage, and pre-existing conditions such as diabetes, vascular disease, and immune deficiencies may be indicative of increased likelihood for developing post surgical complications. Another risk factor of particular interest is the timing of surgery after the incidence of injury. Current literature regarding treatment of hindfoot injuries shows a moderate degree of uniformity, advocating a delay in operative measures until the soft tissue swelling around the injury has had time to subside: a window of approximately 7-14 days after injury. Additionally, in their investigation of Bohler's angle as a predictor for wound healing complications, Shuler and colleagues noted the pre and post operative Bohler's angle differential to be a significant predictor of developing infections, postulating that the increase in heel height during surgery may concomitantly increase soft tissue tension substantially enough to disrupt proper blood supply to the surgical site during healing. These findings lend tremendous support to the idea that blood perfusion in soft tissue plays a significant role in predicting wound healing complications. However, to our knowledge, the use of angiography to correlate pre and post operative soft tissue perfusion patterns with post operative complication in patients undergoing ORIF of fractured calcanei has never been investigated.

Indocyanine green (ICG) angiography has been utilized in a myriad of other fields of medicine to evaluate perfusion in different tissues. It has been used in cardiac surgery to asses bypass patency, in microsurgery to assist in free tissue transfers, and in plastic surgery to assess areas of future necrosis during mastectomy operations. Recently, ICG angiography has been used in general surgery to detect ischemic tissues and aid surgeons in determining the appropriate extent of debridement necessary prior to wound closure in laparotomy procedures. Though its utility in other disciplines of medicine are currently being further developed and understood, the implications of ICG angiography in orthopaedic surgery have gone unrecognized. We postulate that soft-tissue perfusion patterns elucidated by ICG angiography in the heels of patients that have incurred calcaneal fractures may be predictive of wound healing complications that develop after surgery. This information could allow surgeons to greatly reduce the complication rate of open reduction procedures on calcaneus fractures by early utilization of appropriate, patient specific prophylactic measures, and could provide an additional contraindication to this operation for patients whom otherwise were not aware they are at an elevated risk.

ELIGIBILITY:
Inclusion Criteria:

* Persons 18-65 years of age with closed unilateral operative Calcaneus fractures that may be approached by an extended lateral incision

Exclusion Criteria:

* Patients declining participation
* Patients with vascular disease or injury requiring vascular repair
* Patients that have undergone prior ankle or hindfoot surgery
* Patients with additional hindfoot injury or injuries
* Patients with open calcaneal fracture
* Patients with head injury
* Patients with injury greater than 3 weeks old
* Patients who are pregnant or currently nursing
* Patients who are incapable of personally understanding the informed consent document due to mental incapacitation or inability to speak and understand English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Jaeblon, D.O, Principal Investigator — Associate Professor of Orthopaedic Surgery; Associate Director of Orthopaedic Traruma
Locations (1):
- Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Displaced Intra Articular Calcaneus Fracture: displaced intra articular calcaneus fracture with operative repair
Period: Overall Study
Arm/Group | Displaced Intra Articular Calcaneus Fracture
Started | 13
Completed | 0 (Study closed by PI)
Not Completed | 13

BASELINE CHARACTERISTICS:
Groups:
- Operative Calcaneus Fracture: Patients with indications for and electing to undergo operative repair of intra articular calcaneus fracture through extended lateral approach
Arm/Group | Operative Calcaneus Fracture
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Perfusion Data Infection Wound Healing Complication
Description: correlation of multiple absolute and relative data points acquired from near infra red spectroscopy compared to clinical postoperative infection or wound healing complication following lateral approach calcaneus fracture
Time Frame: 3 months postoperative
Population: unable to complete analysis as correlation between clinical and ICG near infra red data acquisition could not be completed do to unexpected lack funding required to pair and analyze extremely large data sets with clinical information as well as too few numbers of patients
Arm/Group | ICG Administered
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Unanticipated Adverse Events Related to ICG: No adverse events related to administration ICG
Arm/Group | Unanticipated Adverse Events Related to ICG
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unanticipated Adverse Events Related to ICG (N=13)
wound healing delay (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes